CLINICAL TRIAL: NCT05693194
Title: Prevalence of Anemia in PICU Survivors: Epidemiology, Pathophysiology and Consequences
Brief Title: Pathophysiology of Anemia in PICU Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Genevieve Du Pont-Thibodeau, Pediatric intensivist, MD, MSc, Associate Clinical Professor, St. Justine's Hospital
Other Study IDs: 2019-2200
Record Dates: First submitted 2019-03-15; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2007, the TRIPICU trial which demonstrated the safety of tolerating anemia in critically ill children through avoidance of unnecessary red cell transfusions. This landmark study led to practice changes and a reduction in the use of red cell transfusion during PICU stay. However, although this restrictive approach appears safe in the acute setting of PICU, there is a paucity of data regarding its long-term impact on the burden of anemia at discharge. Although 98% of patients now survive their PICU stay, we and other groups have documented that around 50% of PICU admissions will be anemic at discharge. A major contributing factor may be the increasing adoption of restrictive red cell transfusion policies during the phase of ICU admission. Given that there are approximately 9000 PICU admissions/year in Canada, this represents almost 4500 children are discharged with anemia.

The causes of anemia are multifactorial, including inflammation, co-morbidities and nutritional, including iron depletion. Anemia, in particular iron deficiency anemia, is well recognized to be associated with abnormal neurocognitive development in infants and young children. Anemia can also contribute to lower exercise tolerance levels impeding children's development and quality of life.

This protocol describes a prospective observational cohort study of PICU survivors, to better understand the epidemiology of anemia at and after PICU discharge. The primary aim will be to determine the prevalence of anemia at 2 months after PICU discharge (primary aim) as well as at 6 and 12 months follow-up (secondary aim). We will evaluate the association of anemia with neurocognitive dysfunction, and quality of life (secondary aim). We will also investigate the pathophysiology of anemia after PICU discharge. We will perform blood tests on anemic patients to measure inflammatory markers as well as markers of iron deficiency (including the new biomarker hepcidin) (tertiary aim).All patients included will be followed while hospitalized in the PICU, as well as at dedicated clinics at 2, 6, and 12 months after PICU discharge.

Anemia affects a large proportion of PICU survivors. This study will allow us to better understand the long-term prevalence and causes of anemia in this population as well as potential association with long-term outcome. Anemia (specifically iron responsive anemia) could be a potentially readily modifiable risk factor, to improve the long-term well-being of these children.

DETAILED DESCRIPTION:
Research Question/Objectives

Primary aim:

1. To determine the prevalence of anemia in PICU survivors at 2 months post PICU discharge. Anemia is defined as per the World Health Organization criteria.

   Hypothesis: Based on the adult literature and our preliminary data, we suspect that at least 30% of children will remain anemic at 2 months after PICU discharge.

   Secondary aims:
2. To determine the prevalence of anemia in PICU survivors at 6 months and 12 months after PICU discharge.
3. To determine the association between post-PICU anemia and neurocognitive outcome at 2, 6, 12 months after PICU discharge.
4. To determine the association of post-PICU anemia with exercise tolerance at 2, 6, 12 months after PICU discharge.
5. To determine the association of post-PICU anemia with quality of life at 2, 6, 12 months after PICU discharge.

   Tertiary aims:
6. To explore the etiology of anemia, by determining the blood levels of iron, transferrin, proportion of transferrin saturation, blood concentration of inflammatory markers - interleukin-6(IL-6), C-reactive protein and erythropoietin (EPO) - and novel markers such as hepcidin - in anemic PICU survivors at PICU discharge, 2,6, and 12 months.
7. To determine the PICU risks factors associated with post-PICU anemia
8. Determine the tolerance and compliance of patients treatment with iron at or after PICU discharge, if prescribed.

Methods We will perform a prospective cohort study of children admitted to the PICU of CHUSJ over a 24-month period. We will include children who: 1) are <18 years; AND 2) have a PICU length of stay at least 4 days; AND 3) required invasive mechanical ventilation ≥ 48 hours. We will exclude patients who underwent cardiac surgery for congenital heart disease, and patients or parents who do not speak English or French. The purpose of these inclusion criteria is to enrol sicker children with significant critical illness and exclude "healthier" children who are admitted to PICU for monitoring and observation (intoxication, post-operative pain management, etc.). Patients with cardiac surgery will be studied in another trial.

This study will include 2 phases: 1) data collection during PICU hospitalization; and 2) follow-up. At CHUSJ, PICU survivors who match our eligibility criteria are currently followed at the PICU follow-up clinic. These patients will be seen and evaluated at 2, 6 and 12 months post-PICU discharge. Research assistants will screen PICU patients daily to identify children with our inclusion criteria. Once patient consent and are enrolled in the study, a research assistant will collect all the clinical variables required for the study and will schedule follow-up appointments upon their discharge.

The primary outcome is the prevalence of anemia at 2 months after PICU discharge. To answer this question, we will measure peripheral blood count, which includes a hemoglobin concentration, in all patients at PICU discharge, and at 2, 6 and 12 months follow-up in patients found to be anemic at PICU discharge. Children that are found to be anemic at PICU discharge will be managed by the PICU medical team responsible. Patients found anemic at PICU follow-up and will be managed by the responsible pediatric intensivist according the Canadian Pediatric Society Guidelines.

To determine the etiology of anemia; albumin, inflammatory markers (IL-6, C-reactive protein), hepcidin and markers of iron status and erythropoiesis (blood ferritin level, serum iron, transferrin saturation, erythropoietin, vitamin B12, folate and reticulocytes) will be measured in all patients at PICU discharge and at 2, 6, and 12 months follow-up for patients found anemic or iron deficient at PICU discharge. Serum hepcidin will be measured by enzyme-linked immunosorbent assay (ELISA) (hepcidin-25 high sensitivity. ELISA, DRG Instruments, Marburg, Germany). Erythropoietin requires 5 ml of blood and consequently will only be sampled in children > 10 kg. All other bloodworks require 3 mL.

Risk factors for anemia will be evaluated by collecting clinical variables and demographic data pertaining to patients' PICU stay. This will include medication prescribed at discharge to correct anemia (iron, erythropoietin and/or red cell transfusion). Presently, there are no standardized guidelines for the treatment of anemia post PICU. Therefore, practitioners will be allowed to choose the treatment strategy they believe in.

Neurocognitive function, physical endurance and quality of life will be evaluated at follow-up appointments. A pediatric intensivist or pediatrician will perform a standardized history and physical exam. In collaboration with a neuropsychologist, they will assess neurocognitive and neurologic clinical outcomes. Neurocognitive impairment will be measured with the Bayley Scales of Infant Development III (1-30 months), Wechsler Preschool and Primary Scale of Intelligence IV (WPPSI) (30mo-7yo), Wechsler Intelligence Scale for Children V (WISC)(7-16 yo) and Wechsler Adult Intelligence Scale IV (WAIS)(16yo and older). Patients and parents will also fill standardized questionnaires that estimate exercise endurance (M-ABC2)and quality of life (Peds-QYL Inventory and Infant Toddler Quality of Life Questionnaire)with the support of our research personnel. If a medical or psychosocial problem is detected during the follow-up, we have ensured the availability of the necessary resources within our hospital to refer patients when necessary (medical specialists, psychologist, physiotherapist, social worker).

Iron tolerance and compliance will be determined during physician encounters at follow-up visits as part of a standardized questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 1) are <18 years; AND 2) have a PICU length of stay at least 4 days; AND 3) required invasive mechanical ventilation ≥ 48 hours

Exclusion Criteria:

we excluded children with 1) pre-existing hematologic disorder causing anemia, including treatment with immunosuppressant or cytotoxic drugs; 2) acute or chronic renal failure requiring renal replacement therapy at time of PICU admission; and 3) postoperative cardiac surgery. The local Institutional Review Board approved this study (#2019-2200).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The purpose of these inclusion criteria is to enrol sicker children with significant critical illness and exclude "healthier" children who are admitted to PICU for monitoring and observation (intoxication, post-operative pain management, etc.).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2019-10-03 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anemia at 2 months post PICU discharge | 2 months
  we will measure peripheral blood count, which includes a hemoglobin concentration, in all patients at PICU discharge and at 2 months follow-up in patients found to be anemic at PICU discharge.

SECONDARY OUTCOMES:
Prevalence of anemia at 6 months and 12 months post PICU discharge | 12 months
  we will measure peripheral blood count, which includes a hemoglobin concentration, in all patients at PICU discharge, and at 2, 6 and 12 months follow-up in patients found to be anemic at PICU discharge.
The association between post-PICU anemia and neurocognitive outcome at 2, 6, 12 months after PICU discharge. | 12 months
  Neurodevelopment will be evaluated at follow-up appointments. A pediatric intensivist or pediatrician will perform a standardized history exam. They will assess neurodevelopment through the Ages and Stages Questionnaire (ASQ). In collaboration with a neuropsychologist, they will assess neurocognitive and neurologic clinical outcomes. Neurocognitive impairment will be measured with the Bayley Scales of Infant Development III (1-30 months), Wechsler Preschool and Primary Scale of Intelligence IV (WPPSI) (30mo-7yo), Wechsler Intelligence Scale for Children V (WISC)(7-16 yo) and Wechsler Adult Intelligence Scale IV (WAIS)(16yo and older).
The association of post-PICU anemia with quality of life at 2, 6, 12 months after PICU discharge. | 12 months
  Patients and parents will fill standardized questionnaires that estimate quality of life (Peds-QYL Inventory and Infant Toddler Quality of Life Questionnaire) with the support of our research personnel
The etiology of anemia, by determining the blood levels of iron, transferrin, proportion of transferrin saturation, blood concentration of inflammatory markers - interleukin-6(IL-6), C-reactive protein and erythropoietin | 12 months
  albumin, inflammatory markers (IL-6, C-reactive protein), hepcidin and markers of iron status and erythropoiesis (blood ferritin level, serum iron, transferrin saturation, erythropoietin, vitamin B12, folate and reticulocytes ) will be measured in all patients at PICU discharge and then at 2, 6, and 12 months follow-up for patients found anemic or iron deficient at PICU discharge. All bloodworks except erythropoietin can be capillary samples measured by micromethod. Erythropoietin requires 5 ml of blood and consequently will only be sampled in children > 10 kg and only at PICU discharge
The PICU risks factors associated with post-PICU anemia | 12 months
  Risk factors for anemia will be evaluated by collecting clinical variables and demographic data pertaining to patients' PICU stay. This will include medication prescribed at discharge to correct anemia (iron, erythropoietin and/or red cell transfusion). Presently, there are no standardized guidelines for the treatment of anemia post PICU. Therefore, practitioners will be allowed to choose the treatment strategy they believe in.
The tolerance and compliance of patients treatment with iron at or after PICU discharge, if prescribed. | 12 months
  Iron tolerance and compliance will be determined during physician encounters at follow-up visits as part of a standardized questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Du Pont-Thibodeau, MD,MSc, Principal Investigator — Centre Hospitalier universitaire Sainte-Justine (CHUSJ)
Locations (1):
- Hopital Ste-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No